CLINICAL TRIAL: NCT03044873
Title: Effect of BMS-986165 on the Pharmacokinetics of Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IM011-015
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Autoimmune Diseases; Inflammatory Diseases
MeSH Terms: conditions — Autoimmune Diseases | interventions — deucravacitinib; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS 986165 and Rosuvastatin (Experimental)
  Interventions: Drug: BMS-986165; Drug: Rosuvastatin

INTERVENTIONS:
Drug: BMS-986165 — Rosuvastatin on Day 1. BMS 986165 on Days 5-8 and Days 10-12. On Day 9, BMS 986165 coadministered with an oral dose of rosuvastatin.
Drug: Rosuvastatin — Rosuvastatin on Day 1. BMS 986165 on Days 5-8 and Days 10-12. On Day 9, BMS 986165 coadministered with an oral dose of rosuvastatin.

SUMMARY:
The study is to assess the effect of coadministration of multiple doses of BMS-986165 on the systemic exposure of rosuvastatin in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Healthy male and female participants (not of childbearing potential) as determined by no clinically significant deviation from normal in medical history, physical exam, ECGs, and clinical laboratory determinations
3. Subjects with body mass index of 18 to 32 kg/m2, inclusive.
4. Women participants must have documented proof that they are not of childbearing potential.
5. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of highly effective contraception for the duration of study treatment(s) plus 5 half-lives of BMS-986165 (4 days) plus 90 days (duration of sperm turnover) for a total of 94 days of post BMS-986165 treatment. In addition, male participants must be willing to refrain from sperm donation during this time.

Exclusion Criteria:

1. History of allergy to BMS-986165, rosuvastatin, or related compounds, of myalgia or rhabdomyolysis while taking rosuvastatin or related compounds or any other drug allergy
2. Any significant acute or chronic medical illness, active TB requiring treatment or documented latent TB within the previous 3 years, current or recent gastrointestinal disease, current or recent history of nausea, vomiting, constipation or irregular bowel movement
3. History of chronic headaches, syncope, orthostatic instability, or recurrent dizziness, biliary disorders, drug-induced acne or rash, fibromyalgia, neutropenia or thrombocytopenia
4. Smokers who currently smoke, recent drug or alcohol abuse, blood transfusion within 4 weeks of study treatment administration, current skin findings that could interfere with the interpretation of study

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum observed plasma concentration) of Rosuvastatin. | Up to Day 13
  Measured by plasma concentration.
AUC(0-T) (Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration) of Rosuvastatin. | Up to Day 13
  Measured by plasma concentration.
AUC(INF) (Area under the plasma concentration-time curve from time zero extrapolated to infinite time) of Rosuvastatin. | Up to Day 13
  Measured by plasma concentration.

SECONDARY OUTCOMES:
Number of Subjects with Deaths. | Up till 30 days after discontinuation
  Measured by investigator assessment.
Number of Subjects with Serious Adverse Events. | Up till 30 days after discontinuation
  Measured by investigator assessment.
Number of Subjects with Adverse Events. | Up till 30 days after discontinuation
  Measured by investigator assessment.
Number of subjects with Adverse Events Leading to Discontinuation. | Up till 30 days after discontinuation
  Measured by investigator assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx